CLINICAL TRIAL: NCT05140434
Title: Evaluation of the Predictive Power of Double-product Increase Measured During an Exercise Test for the Prediction of Coronary Stenosis As Diagnosed by Cardiac CT Scan or Coronary Angiography.
Brief Title: Evaluation of the Benefit of Exercise Testing for the Diagnosis of Obstruction in the Coronary Arteries of the Heart
Acronym: DP-Cor-1
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0054
Record Dates: First submitted 2021-11-19; First posted 2021-12-01 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Coronary Artery Disease
Keywords: Exercise testing; coronary stenosis; double product
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Exercise test — exercise test on an exercise bike with increasing load
Diagnostic Test: Cardiac CT — cardiac CT scan

SUMMARY:
The purpose of this study is to determine whether exercise testing can detect an obstruction in a coronary artery, and, thereby, can avoid performing a coronary imaging in some cases.

Patients with a suspicion of coronary artery disease perform an exercise test on an exercise bike with increasing load. EKG, blood pressure, and other parameters are monitored. Patients benefit also of either a cardiac CT scan or a coronary angiography to establish whether they really have coronary obstruction.

DETAILED DESCRIPTION:
Double product DP (product of systolic blood pressure and heart rate) is directly related to the myocardial oxygen consumption (MVO2). Since O2 extraction by the myocyte in maximal at rest, only an increase in coronary blood flow can increase MVO2 during exercise. Therefore, if a coronary stenosis limits the maximal coronary flow, it will limit MVO2 and DP at exercise.

Patients with both an exercise test and a coronary artery imaging (cardiac CT or coronary angiography) within 3 months, are included. DP increase (DP max/DP at rest) is measured during a maximal, symptom-limited exercise on a cycloergometer. DP at rest is measured either before the exercise test, at the end of the recovery period or during a visit to the cardiologist in the 2 months of the test, whichever is the smallest.

The predictive power to detect a significant coronary artery stenosis is assessed by computing a Receiving Operating Characteristic (ROC) curve, its area under the curve, sensitivity, specificity, and decision thresholds.

Number expected: 100-120 Time period of data collection: 1/1/2019 to 3/1/2022

ELIGIBILITY:
Inclusion Criteria:

* Starting betweew 1/1/2019 and 3/1/2022
* 18 year-old patients or older
* Patients with both exercise testing and either Cardiac CT or coronary angiography within 3 months
* Patients informed and not opposing to their participation to the study

Exclusion Criteria:

* Patients unable to fully understand the information related to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out-patients attending Centre Hospitalier Sud Francilien's cardiology department.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2022-05-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area Under the ROC curve | at 3 months
  AUC of the ROC curve defined by DP increase and significant coronary artery stenosis or not

SECONDARY OUTCOMES:
Youden threshold | at 3 months
  Maximalization of the difference between sensitivity and 1-specificity
ROC for women | at 3 months
  AUC for women

CONTACTS AND LOCATIONS:
Overall Officials: Olivier CHARANSONNEY, MD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- CHARANSONNEY Olivier, Corbeil-Essonnes, France, France

IPD SHARING:
Plan to Share IPD: No